CLINICAL TRIAL: NCT01680367
Title: A Comparative Study of Dressings for Split-Thickness Skin Graft Donor Sites.
Brief Title: Wound Dressings For Split-Thickness Skin Graft Donor Sites in Patients Undergoing Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OSU-06043; NCI-2012-00985 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-09-04; First posted 2012-09-07 (Estimated); Last update posted 2016-03-18 (Estimated); Status verified 2016-03

CONDITIONS: Pain; Perioperative/Postoperative Complications
MeSH Terms: conditions — Pain; Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (control) (Experimental): Patients receive transparent film dressing (otolaryngology service) or Xeroform petroleum gel impregnated gauze dressing (surgical oncology service) after surgery.
  Interventions: Procedure: wound care management; Other: questionnaire administration
- Arm II (native collagen wound dressing) (Experimental): Patients receive native collagen wound dressing after surgery.
  Interventions: Procedure: wound care management; Other: questionnaire administration

INTERVENTIONS:
Procedure: wound care management — Receive transparent film dressing or Xeroform petroleum gel impregnated gauze dressing
  Arms: Arm I (control)
Procedure: wound care management — Receive native collagen wound dressing
  Arms: Arm II (native collagen wound dressing)
Other: questionnaire administration — Ancillary studies

SUMMARY:
This study is to determine what dressing would work best to heal and keep from hurting, the split-thickness skin graft donor site which will be done as part of the patient's surgical procedure. Currently there is a dressing that is transparent and it is placed on the wound after surgery and wrapped with gauze and an elastic bandage. Two days after the surgery the gauze and elastic bandages are removed and the area is left with the transparent dressing. Sometimes the dressing needs to be changed because it leaks. On the fifth day this dressing is removed and the wound is left open to air. The dressing researchers are studying is a dressing that has been used for different types of wounds, as well as this type of wound. It is applied in the same manner; however, it is left in place until it falls off independently, usually around post-operative (post-op) day 10.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Which dressing type and technique is most effective in minimizing pain and inflammation and promoting epithelialization in patients who have had surgery which requires the use of an anterior thigh split-thickness skin graft?

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive transparent film dressing (otolaryngology service) or Xeroform petroleum gel impregnated gauze dressing (surgical oncology service) after surgery.

ARM II: Patients receive native collagen wound dressing after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Population of otolaryngological or surgical oncology patients experiencing an autologous split-thickness skin graft as part of their surgical procedure
* Patients will have a Glasgow Coma score of 15 (or 10 with a tracheostomy)
* Patient donor sites will be limited to the anterior thigh
* Patients will be free of documented circulatory deficits, neuropathy, or mental illness which prohibits their ability to independently consent or respond to questions regarding pain
* Patients will be able to give consent independently
* Patients will be able to read and write in English

Exclusion Criteria:

* Patients unable to give independent consent for any reason
* Skin graft donor sites other than the anterior thigh
* Patients with a concurrent diagnosis of diabetes, peripheral vascular disease, and/or paresthesias or paralysis of the lower extremities
* Patients who are unable to complete a self-report pain scale
* Patients who are prisoners
* Patients who are known active alcoholics
* Patients on steroids or other medications known to affect healing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2008-11; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Pain score ranging in value from 0 to 10 | Up to 14 days
  Initial analyses will include two sample t-tests (or a nonparametric equivalent, if more appropriate) for each day to compare the mean pain scores for each treatment group. The pain score will be evaluated using multiple linear regression, while multiple logistic or polytomous regression will be used for the categorical outcomes.

SECONDARY OUTCOMES:
Distress checklist score | Up to 14 days
  The specific modeling approach for the distress score will depend on the range of values obtained. Standard model building techniques will be employed and clinically important interactions between covariates and the groups will be explored.
Inflammation as measured by the Wound Assessment Inventory (WAI) | Up to 14 days
Categorical epithelialization assessment | Up to 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hofacre, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu